CLINICAL TRIAL: NCT06163456
Title: Influence of Cardiorespiratory Fitness and Body Composition on Resting and Post-exercise Indices of Vascular Health in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Towson University (Other)
Responsible Party: Principal Investigator, Rian Q. Landers-Ramos, Assistant Professor, Towson University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1810041426
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Endothelial Dysfunction; Arterial Stiffness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- low fitness (Experimental)
  Interventions: Other: Acute submaximal exercise
- moderate fitness (Active Comparator)
  Interventions: Other: Acute submaximal exercise
- high fitness (Active Comparator)
  Interventions: Other: Acute submaximal exercise

INTERVENTIONS:
Other: Acute submaximal exercise — 30 min of treadmill running at 70% of the participants maximal oxygen consumption

SUMMARY:
This research is being done to determine whether acute exercise causes differences in numbers of novel blood factors associated with vascular health in college-aged adults across different physical activity habits. As only ~50% of cardiovascular (CV) events can be explained by traditional CV risk factors such as high blood pressure and high cholesterol, it is anticipated that this research will provide a more comprehensive look into novel risk factors that may better explain CV risk and that may be modifiable through regular physical activity.

ELIGIBILITY:
Inclusion Criteria:

* 18-29 years of age; healthy male and female; Physically inactive, defined as participation in less than 20 min of continuous endurance exercise on fewer than 2 days/week; Recreationally active, defined as participation in 30 min/day of moderate-intensity cardiovascular activity on greater than 4 days/week; Highly active- defined as performing 30-60 min of moderate- to vigorous-intensity endurance exercise greater than 5 days/week.

Exclusion Criteria:

* currently pregnant, previously diagnosed coronary heart disease or congenital heart disease, serum total cholesterol >200 mg/dl, low-density lipoprotein cholesterol >130 mg/dl, high-density lipoprotein cholesterol < 35 mg/dl, fasting glucose >100 mg/dl, systolic blood pressure > 130 mmHg, diastolic blood pressure >90 mmHg, and BMI >30 kg/m2.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
endothelial function | Baseline and 60 min post-exercise
  flow-mediated dilation
arterial stiffness | Baseline and 60 min post-exercise
  augmentation index

CONTACTS AND LOCATIONS:
Overall Officials: Rian Q Landers-Ramos, PhD, Principal Investigator — Towson University
Locations (1):
- Towson University, Towson, Maryland, United States

IPD SHARING:
Plan to Share IPD: No